CLINICAL TRIAL: NCT03027427
Title: Prospective Evaluation and Molecular Profiling in Patients With Gastric Tumors
Brief Title: Prospective Evaluation and Molecular Profiling in People With Gastric Tumors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170044; 17-C-0044
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Stomach Neoplasms; Stomach Cancer
Keywords: Screening; Heritable Gastric Malignancy; Molecular Profiling; Molecular Alterations
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with confirmation of, or suspicion of, a heritable gastric malignancy disorder

SUMMARY:
Background:

Certain stomach cancers are rare, but they have high mortality rates. Researchers want to learn more about gastric (stomach) tumors. In this study, they want to collect data from people who have stomach cancer or are at risk to get it. This data will be used to see if the people can be in other studies.

Objective:

To study tissue from stomach tumors and find people eligible for more studies on gastric cancer.

Eligibility:

Age greater than or equal to 2 years old who have or may have stomach cancer, lesions that may be related to stomach cancer, or an inherited disorder that leads to stomach cancer.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Heart tests

Scans or ultrasound.

For the scans, participants lie in a machine that takes pictures. For some scans, they will swallow or be injected with a small amount of radioactive material. Special cameras will show the material in the body.

Tumor sample taken with a needle or surgery

Some participants will have an endoscopy. A long, flexible tube with a camera will be inserted through the mouth into the stomach. The tube will collect tissue from the stomach.

Some participants may have follow-up visits. Some may be invited to join other studies. Others will be contacted by phone to see how they are doing.

...

DETAILED DESCRIPTION:
Background:

* Greater than 90% of gastric tumors are of epithelial origin and are classified as adenocarcinomas; the remainders include GIST, carcinoid and lymphoma.
* Gastric adenocarcinoma is rare in the United States (incidence 7.4 per 100,000).
* Mortality rates are high with an estimated 5-year overall survival of 25% - 30%.
* Up to 3% of gastric adenocarcinomas occur as part of a heritable cancer syndrome.
* Molecular sub-classification of gastric adenocarcinomas has been reported, however translation of these findings into clinical management of patients has yet to occur.

Objectives:

* To permit clinical and laboratory evaluation and molecular profiling of tumor tissue from patients with gastric malignancies or non-invasive (neoplastic) conditions.
* Assess eligibility for enrollment in studies of gastric cancer conducted in the CCR.
* To allow long-term follow up of patients with gastric tumors, or heritable gastric malignancy syndromes, to support clinical and preclinical research particularly related to molecular alterations in gastric tumors and their response to therapy.

Eligibility:

Patients with any of the following are eligible:

* Malignant or non-invasive, neoplastic lesions of the stomach confirmed by histopathology or cytopathology;
* Suspicious lesions not yet confirmed, but considered likely related to the stomach pending further evaluation;
* Confirmed, deleterious germline mutation (including but not limited to HDGC, GAPPS) known to predispose to gastric tumors;
* Confirmed or suspicious heritable gastric malignancy disorder;
* Clinically suspicious personal or family medical history of gastric cancer or gastric cancer syndrome that warrants genetics evaluation.
* Age greater than or equal to 2 years.

Design:

* This protocol is designed to facilitate clinical evaluation, molecular tumor profiling, and long-term follow up of patients with gastric tumors.
* Patients will be screened and clinical evaluation performed to determine eligibility for other CCR trials for gastric tumors.
* No investigational treatment will be administered and no procedures will be done for only research purposes on this protocol.
* It is anticipated that the protocol will enroll a maximum of 250 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with any of the following are eligible:

  * Malignant or non-invasive, neoplastic lesions of the stomach confirmed by histopathology or cytopathology in a CLIA-certified laboratory;
  * Suspicious lesions not yet confirmed, but considered likely to be related to the stomach pending further evaluation;
  * Confirmed, deleterious germline mutation (including but not limited to HDGC, GAPPS) known to predispose to gastric tumors;
  * Confirmed or suspicious heritable gastric malignancy disorder;
  * Clinically suspicious personal or family medical history of gastric cancer or gastric cancer syndrome that warrants genetics evaluation.
* Patients must have an ECOG performance score of 0-2.
* Age greater than or equal to 2 years. Note: Patients greater than or equal to 2 and less than or equal to 18 years of age may only participate in research sample collection if the tissue acquisition is performed during a clinically indicated surgical procedure, and the sampling of tissue, blood and urine does not add risk to the clinically indicated procedures.
* The patient is a candidate for the clinically indicated medical evaluations that are being offered
* Ability of subject, their parents/guardians or legally authorized representative (LAR) to understand and must be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

Candidates who do not meet the inclusion criteria.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmation of, or suspicion of, a heritable gastric malignancy disorder
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Long-term follow up to support clinical and preclinical research | follow up
  long-term follow up of patients with gastric tumors, or heritable gastric malignancy syndromes screened on this study, to support clinical and preclinical research particularly related to molecular alterations in gastric tumors and their response to therapy
Determination of eligibility | at initial visit
  determination of eligibility for enrollment in studies of gastric cancer conducted in the CCR
Clinical and laboratory evaluation and molecular profiling of tumor tissue | at initial visit and as clinically indicated
  Tissue samples collected to permit clinical and laboratory evaluation and molecular profiling of tumor tissue from patients with gastric malignancies or non-invasive (neoplastic) conditions

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Blakely, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Wang K, Yuen ST, Xu J, Lee SP, Yan HH, Shi ST, Siu HC, Deng S, Chu KM, Law S, Chan KH, Chan AS, Tsui WY, Ho SL, Chan AK, Man JL, Foglizzo V, Ng MK, Chan AS, Ching YP, Cheng GH, Xie T, Fernandez J, Li VS, Clevers H, Rejto PA, Mao M, Leung SY. Whole-genome sequencing and comprehensive molecular profiling identify new driver mutations in gastric cancer. Nat Genet. 2014 Jun;46(6):573-82. doi: 10.1038/ng.2983. Epub 2014 May 11. PMID 24816253
- [Background] Cristescu R, Lee J, Nebozhyn M, Kim KM, Ting JC, Wong SS, Liu J, Yue YG, Wang J, Yu K, Ye XS, Do IG, Liu S, Gong L, Fu J, Jin JG, Choi MG, Sohn TS, Lee JH, Bae JM, Kim ST, Park SH, Sohn I, Jung SH, Tan P, Chen R, Hardwick J, Kang WK, Ayers M, Hongyue D, Reinhard C, Loboda A, Kim S, Aggarwal A. Molecular analysis of gastric cancer identifies subtypes associated with distinct clinical outcomes. Nat Med. 2015 May;21(5):449-56. doi: 10.1038/nm.3850. Epub 2015 Apr 20. PMID 25894828
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of gastric adenocarcinoma. Nature. 2014 Sep 11;513(7517):202-9. doi: 10.1038/nature13480. Epub 2014 Jul 23. PMID 25079317
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0044.html